CLINICAL TRIAL: NCT00176618
Title: The Effects of Curcuminoids on Aberrant Crypt Foci in the Human Colon
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: principal Investigator left institution
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: C. S. Yang, PhD, The Cancer Institute of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4611; CINJ#120305
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Aberrant Crypt Foci
Keywords: Aberrant Crypt Foci
MeSH Terms: conditions — Aberrant Crypt Foci | interventions — Sulindac; Curcumin

INTERVENTIONS:
Drug: sulindac — Sulindac 150 mg po BID
Drug: curcumin — Curcumin 250 mg po BID

SUMMARY:
The purpose of this study is to determine the effectiveness of curcumin in reducing the number of aberrant crypt foci (ACF) in the colon.

DETAILED DESCRIPTION:
Laboratory studies have indicated that this agent, which is derived from plants and found in foods we eat, has anti-inflammatory properties and prevents colon cancer in animal studies. ACFs are small abnormalities in the lining of the colon that with time may grow into colorectal adenomas (also called polyps, growths or small masses of tissue on the lining of the colon or rectum which have the potential to become cancerous) which can then grow into adenocarcinomas (cancer) in the colon or rectum.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be eligible for colorectal cancer (CRC) screening/surveillance by current criteria.
* Subjects must have at least 5 ACF on eligibility chromosigmoidoscopy examination.

Exclusion Criteria:

Subjects must not have:

* Alcohol consumption of greater than 2 glasses of wine or beer per day or illicit recreational drug use
* Platelet or coagulation abnormalities, or personal history of a bleeding disorder, including individuals taking warfarin.
* High risk for developing endocarditis (history of endocarditis or rheumatic fever, cardiac valve prostheses, or mitral valve prolapse that requires antibiotic prophylaxis).
* Uncontrolled hypertension, diabetes, or chronic congestive heart failure.
* Renal insufficiency defined as a serum creatinine > 2.5 mg/dl
* History of colorectal surgery with removal of the distal 60 cm of colon or rectum.
* History of other gastrointestinal mucosal epithelial diseases (such as Barrett's esophagus, chronic or recurrent peptic ulcer disease, celiac sprue or other disorders of nutrient absorption).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of curcumin or the NSAID sulindac on the number of ACF in the left colon and rectum of normal volunteers found to have them on an initial magnifying chromoendoscopic screening exam | 48 months

SECONDARY OUTCOMES:
To determine the turnover (proliferation, apoptosis, and differentiation) of colorectal epithelial cells in the crypts in situ in response to each treatment | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Yang CS, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States